CLINICAL TRIAL: NCT03647020
Title: Impact of Oocytes With CLCG on ICSI Outcomes and Their Potential Relation to Pesticide Exposure
Acronym: CLCG-ICSI
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2017_843_0044
Record Dates: First submitted 2018-08-23; First posted 2018-08-27 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2018-08

CONDITIONS: Pesticide Poisoning
Keywords: oocyte; ovarian stimulation; dysmorphic cytoplasm

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Oocyte quality is a key limiting factor in female fertility which is primarily reflected in morphological features. Centrally located cytoplasm granulation (CLCG) is one type of cytoplasmic dimorphism exhibited by oocytes that could be linked to pesticide exposure with a significant risk of decreased ICSI outcomes.

This retrospective study included 633 women who were part of an intracytoplasmic spermatozoa injection (ICSI) program between 2009 and 2011. The participants lived in the Picardy region of France and had been exposed to pesticides. The participants were divided in two groups based on prevalence of oocytes with CLCG (LCLCG [n= 83]: low prevalence of oocytes with CLCG under 25%. HCLCG [ n= 68]: high prevalence of CLCG over 75%). The embryological and clinical outcomes were analysed for both groups and were calculated using the difference between the two values.

DETAILED DESCRIPTION:
Oocyte quality is a key limiting factor in female fertility which is primarily reflected in morphological features. Centrally located cytoplasm granulation (CLCG) is one type of cytoplasmic dimorphism exhibited by oocytes that could be linked to pesticide exposure with a significant risk of decreased ICSI outcomes.

This retrospective study included 633 women who were part of an intracytoplasmic spermatozoa injection (ICSI) program between 2009 and 2011. The participants lived in the Picardy region of France and had been exposed to pesticides. The participants were divided in two groups based on prevalence of oocytes with CLCG (LCLCG [n= 83]: low prevalence of oocytes with CLCG under 25%. HCLCG [ n= 68]: high prevalence of CLCG over 75%). The embryological and clinical outcomes were analysed for both groups and were calculated using the difference between the two values. The included population in the investigator's retrospective study consisted of 633 couples who attended a reproductive medical center and who were part of an ICSI program between 2009 and 2011.

ELIGIBILITY:
Inclusion Criteria:

* couples who attendes a reproductive medical center
* couples that were part of a ICSI program between 2009 and 2011
* women were normo-responders
* female > 18 years <35 yeas old

Exclusion Criteria:

* female < 18 years > 35 yeas old
* couple with severe male infertility factors on oocyte activation and subsequent embryo development

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population in the retrospective study consisted of 633 couples who attended a reproductive medical center and who were part of an ICSI program between 2009 and 2011. The study population is described in Table
  1. In the selected couples, women were normo-responders (oocyte cohort over 5), under 35 years old, living in the Picardy, France region, and exhibited CLCG after oocyte morphology evaluation which was confirmed by a second embryologist (Fig. 1
Sampling Method: Probability Sample
Enrollment: 633 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2017-06-06 (Actual); Study Completion 2017-06-06 (Actual)

PRIMARY OUTCOMES:
ICS outcomes of couples presenting differetn CLCG prevalence | 2years
  The aim of the present study was to investigate the ICSI outcomes of couples presenting different CLCG prevalence's of retrieved oocytes (low prevalence of CLCG; fewer than 25% [LCLCG] and high prevalence of CLCG; over 75% [HCLCG]) and its correlation to pesticide exposure zones in the region of Picardy, France.

CONTACTS AND LOCATIONS:
Overall Officials: Moncef Ben Khlifa, MD, Principal Investigator — CHU AMIENS

IPD SHARING:
Plan to Share IPD: No